CLINICAL TRIAL: NCT01922349
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses and Multiple Rising Oral Doses of BI 113608 in Healthy Male Asian and Caucasian Volunteers (Randomised, Double-blind, Placebo-controlled Within Dose Groups)
Brief Title: Safety, Tolerability and Pharmacokinetics of BI 113608 in Healthy Asian and Caucasian Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1314.9
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (8):
- Placebo (Multiple dose) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Dose 1, Single dose (Experimental): Low dose
  Interventions: Drug: BI 113608
- Dose 2, Single dose (Experimental): Medium dose
  Interventions: Drug: BI 113608
- Dose 3, Single dose (Experimental): High dose
  Interventions: Drug: BI 113608
- Dose 4, Multiple dose (Experimental): Low dose
  Interventions: Drug: BI 113608
- Dose 5, Multiple dose (Experimental): Medium dose
  Interventions: Drug: BI 113608
- Dose 6, Multiple dose (Experimental): High dose
  Interventions: Drug: BI 113608
- Placebo (Single dose) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 113608 — Medium dose (Multiple dosing)
  Arms: Dose 5, Multiple dose
Drug: Placebo — Placebo (Multiple dosing)
  Arms: Placebo (Multiple dose)
Drug: BI 113608 — Low dose (Multiple dosing)
  Arms: Dose 4, Multiple dose
Drug: Placebo — Placebo (Single dosing)
  Arms: Placebo (Single dose)
Drug: BI 113608 — High dose (Single dosing)
  Arms: Dose 3, Single dose
Drug: BI 113608 — Medium dose (Single dosing)
  Arms: Dose 2, Single dose
Drug: BI 113608 — Low dose (Single dosing)
  Arms: Dose 1, Single dose
Drug: BI 113608 — High dose (Multiple dosing)
  Arms: Dose 6, Multiple dose

SUMMARY:
Safety, tolerability and pharmacokinetics of single and multiple oral doses of BI 113608 in healthy Chinese, Japanese and Caucasian male volunteers.

ELIGIBILITY:
Inclusion criteria:

-Healthy male volunteers according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure, Pulse Rate), 12-lead Electrocardiogram, clinical laboratory tests

* Chinese ethnicity, Japanese ethnicity according to the following criteria Japanese; born in Japan, be a current Japanese passport holder, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan Chinese; ethnic Chinese, born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China
* Caucasian
* Age older than 20 and younger than 45 years
* Normal lung function testing
* Normal peripheral oxygen saturation as determined by non-invasive pulse oxymetry
* Body Mass Index more than 18.5 and Body Mass Index less than 25 kg/m2 for Japanese and Chinese
* Body Mass Index more than 18.5 and Body Mass Index less than 29.9 kg/m2 for Caucasians
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation.

Exclusion criteria:

* Any finding of the medical examination (including Blood Pressure, Pulse Rate and Electrocardiogram) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (including but not limited to any kind of seizures, migraine, stroke or psychiatric disorders) within the past 6 month
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 20 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
* A history of additional risk factors for Torsades de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1314.9.8201 Boehringer Ingelheim Investigational Site, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo tablet: oral administration, single dose (single rising dose(SRD) period) followed by twice a day for 13 days plus a single dose on day 14 (Multiple rising dose (MRD) period)
- BI 113608 - 10 mg: 2 conventional tablets 5 mg BI 113608 oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period)
- BI 113608 - 25 mg: 1 conventional tablet 25 mg BI 113608 oral administration, once daily (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period)
- BI 113608 - 50 mg: 2 conventional tablets 25 mg BI 113608 oral administration, once daily (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period)
Period: Single Rising Dose (SRD) Period
Arm/Group | Placebo | BI 113608 - 10 mg | BI 113608 - 25 mg | BI 113608 - 50 mg
Started | 25 | 27 | 18 | 27
Completed | 25 | 27 | 18 | 27
Not Completed | 0 | 0 | 0 | 0
Period: Multiple Rising Dose (MRD) Period
Arm/Group | Placebo | BI 113608 - 10 mg | BI 113608 - 25 mg | BI 113608 - 50 mg
Started | 24 (One subject discontinued the trial after the SRD period due to non-compliance with the protocol.) | 27 | 18 | 27
Completed | 24 | 27 | 18 | 26
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all subjects who were dispensed trial medication and were documented to have taken at least 1 dose of the investigational treatment.
Groups:
- Placebo: Matching placebo tablet: oral administration, single dose (single rising dose(SRD) period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period)
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 113608 - 10 mg | BI 113608 - 25 mg | BI 113608 - 50 mg | Total
Number analyzed (Participants) | 25 | 27 | 18 | 27 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (5.1) | 28.5 (4.4) | 28.3 (6.4) | 28.5 (5.2) | 28.3 (5.2)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 25 | 27 | 18 | 27 | 97

OUTCOME MEASURES:

1. Primary Outcome: Number (%) of Subjects With Drug-related Adverse Events
Description: Percentage of subjects with drug-related adverse events (AE) in the SRD and MRD periods combined. The investigator assessed the possible causal relationship between an AE and the trial medication.
Time Frame: Up to 21 days (4 days for SRD period and 17 days for MRD period)
Population: Treated set (TS)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BI 113608 - 10 mg | BI 113608 - 25 mg | BI 113608 - 50 mg
Number analyzed (Participants) | 25 | 27 | 18 | 27
Percentage of participants | 28.0 | 51.9 | 33.3 | 92.6

2. Secondary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma)
Description: maximum measured concentration of the analyte in plasma after a single dose of BI 113608.
Time Frame: 0.25 hours (h), 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 36h, 48h, 71.75h after drug administration
Population: The PK analysis set (PKS) included all subjects of the TS who provided at least 1 secondary PK endpoint in any dose period, which was judged as PK evaluable and was not affected by important protocol violation(s) relevant to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- BI 113608 - 10 mg - Chinese: 2 conventional tablets 5 mg BI 113608 orally administered single dose in Chinese subjects (SRD period)
- BI 113608 - 10 mg - Japanese: 2 conventional tablets 5 mg BI 113608 orally administered single dose in Japanese subjects (SRD period)
- BI 113608 - 10 mg - Caucasian: 2 conventional tablets 5 mg BI 113608 orally administered single dose in Caucasian subjects (SRD period)
- BI 113608 - 25 mg - Chinese: 1 conventional tablet 25 mg BI 113608 orally administered single dose in Chinese subjects (SRD period)
- BI 113608 - 25 mg - Japanese: 1 conventional tablet 25 mg BI 113608 orally administered single dose in Japanese subjects (SRD period)
- BI 113608 - 50 mg - Chinese: 2 conventional tablets 25 mg BI 113608 orally administered single dose in Chinese subjects (SRD period)
- BI 113608 - 50 mg - Japanese: 2 conventional tablets 25 mg BI 113608 orally administered single dose in Japanese subjects (SRD period)
- BI 113608 - 50 mg - Caucasian: 2 conventional tablets 25 mg BI 113608 orally administered single dose in Caucasian subjects (SRD period)
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
nmol/L | 45.8 (71.4) | 72.7 (63.6) | 38.9 (40.1) | 191 (55.8) | 217 (37.2) | 494 (36.8) | 320 (71.4) | 437 (28.7)

3. Secondary Outcome: Tmax (Time From Dosing to Maximum Measured Concentration in Plasma)
Description: Time from dosing to maximum measured concentration in plasma after a single dose of BI 113608.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
hour | 1.00 [0.500 to 4.00] | 0.75 [0.50 to 4.00] | 0.75 [0.50 to 2.00] | 0.50 [0.25 to 3.00] | 0.75 [0.50 to 1.50] | 0.50 [0.50 to 4.00] | 0.75 [0.50 to 2.50] | 0.75 [0.50 to 1.00]

4. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after a single dose of BI 113608.
Time Frame: 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 36h, 48h, 71.75h after drug administration
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
nmol*h/L | 199 (39.6) | 288 (26.8) | 196 (20.1) | 648 (29.9) | 775 (28.7) | 1560 (23.1) | 1320 (48.7) | 1410 (21.0)

5. Secondary Outcome: AUC0-tz (Area Under the Concentration-time Curve of the Analyte in Plasma From Time 0 to Time of Last Quantifiable Data Point)
Description: Area under the concentration-time curve of the analyte in plasma from time 0 to time of last quantifiable data point after a single dose of BI 113608.
Time Frame: 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 36h, 48h, 71.75h after drug administration
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
nmol*h/L | 197 (39.9) | 285 (27.2) | 193 (19.8) | 645 (30.4) | 773 (28.7) | 1560 (23.2) | 1320 (48.9) | 1400 (20.9)

6. Secondary Outcome: t1/2 (Terminal Half-life of the Analyte in Plasma After the First Dose)
Description: Terminal half-life of the analyte in plasma after a single dose of BI 113608.
Time Frame: 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 36h, 48h, 71.75h after drug administration
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
hours | 12.7 (45.0) | 12.1 (29.3) | 15.4 (33.2) | 11.7 (29.8) | 10.1 (23.0) | 11.7 (18.2) | 10.7 (15.3) | 12.9 (21.8)

7. Secondary Outcome: Cmax,ss
Description: Maximum measured concentration of the analyte in plasma at steady state
Time Frame: 23.92h, 71.92h, 119.92h, 167.92h, 215.92h, 227.92h, 263.92h, 275.92h, 311.92h, 312.25h, 312.5h, 312.75h, 313h, 313.5h, 314h, 314.5h, 315h, 316h, 318h, 320h, 322h, 324h, 328h, 336h, 348h, 360h, 384h
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- BI 113608 - 10 mg - Chinese: 2 conventional tablets 5 mg BI 113608 oral administration twice a day for 13 days plus a single dose on day 14 in Chinese subjects (MRD period)
- BI 113608 - 10 mg - Japanese: 2 conventional tablets 5 mg BI 113608 oral administration twice a day for 13 days plus a single dose on day 14 in Japanese subjects (MRD period)
- BI 113608 - 10 mg - Caucasian: 2 conventional tablets 5 mg BI 113608 oral administration twice a day for 13 days plus a single dose on day 14 in Caucasian subjects (MRD period)
- BI 113608 - 25 mg - Chinese: 1 conventional tablet 25 mg BI 113608 oral administration twice a day for 13 days plus a single dose on day 14 in Chinese subjects (MRD period)
- BI 113608 - 25 mg - Japanese: 1 conventional tablet 25 mg BI 113608 oral administration twice a day for 13 days plus a single dose on day 14 in Japanese subjects (MRD period)
- BI 113608 - 50 mg - Chinese: 2 conventional tablets 25 mg BI 113608 oral administration twice a day for 13 days plus a single dose on day 14 in Chinese subjects (MRD period)
- BI 113608 - 50 mg - Japanese: 2 conventional tablets 25 mg BI 113608 oral administration twice a day for 13 days plus a single dose on day 14 in Japanese subjects (MRD period)
- BI 113608 - 50 mg - Caucasian: 2 conventional tablets 25 mg BI 113608 oral administration twice a day for 13 days plus a single dose on day 14 in Caucasian subjects (MRD period)
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 9
nmol/L | 42.5 (66.4) | 66.5 (54.1) | 33.7 (48.2) | 223 (56.7) | 234 (33.2) | 500 (19.0) | 409 (43.2) | 407 (27.0)

8. Secondary Outcome: Tmax,ss
Description: Time from last dosing to maximum concentration of the analyte in plasma at steady state
Time Frame: as for outcome 7
Population: PKS
Measure: Median (Full Range); unit: hours
Groups:
- BI 113608 - 10 mg - Chinese: 2 conventional tablets 5 mg BI 113608 oral administration twice a day for 13 days plus a single dose on day 14 days in Chinese subjects (MRD period)
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 9
hours | 0.75 [0.50 to 6.00] | 0.75 [0.50 to 3.00] | 1.00 [0.50 to 4.00] | 0.75 [0.25 to 3.00] | 0.75 [0.50 to 1.50] | 0.75 [0.50 to 1.50] | 0.767 [0.75 to 4.00] | 0.75 [0.50 to 3.00]

9. Secondary Outcome: AUCtau,ss
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval tau
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 9
nmol*h/L | 222 (26.9) | 273 (35.7) | 199 (31.7) | 860 (33.4) | 823 (20.5) | 2000 (6.46) | 1560 (22.0) | 1530 (41.5)

10. Secondary Outcome: t1/2,ss
Description: Terminal half-life of the analyte in plasma at steady state
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 9
hours | 13.6 (10.4) | 15.3 (25.1) | 16.6 (51.0) | 13.2 (23.3) | 13.1 (9.43) | 13.4 (16.8) | 12.4 (6.97) | 13.7 (35.8)

11. Secondary Outcome: RA,Cmax (Accumulation Ratio of the Analyte in Plasma at Steady State After Multiple Oral Administration Over a Uniform Dosing Interval Tau)
Description: Accumulation ratio of the analyte in plasma at steady state after multiple oral administration over a uniform dosing interval tau, expressed as ratio of Cmax at steady state and after single dose
Time Frame: 0.25h,0.5h,0.75h,1h,1.5h,2h,2.5h,3h,4h,6h,8h,10h,12h,16h,24h,36h,48h,~72h in SRD and ~24h,~72h,~120h,~168h,~216h,~228h,~264h,~276h,~312h,~312.25h,312.5h,312.75h,313h,313.5h,314h,314.5h,315h,316h,318h,320h,322h,324h,328h,336h,348h,360h,384h in MRD
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Cmax
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 9
Ratio of Cmax | 0.928 (52.2) | 0.915 (31.4) | 0.866 (34.1) | 1.17 (61.2) | 1.08 (37.2) | 1.01 (23.6) | 1.39 (64.4) | 0.931 (36.1)

12. Secondary Outcome: RA,AUC (Accumulation Ratio of the Analyte in Plasma at Steady State After Multiple Dose Administration Over a Uniform Dosing Interval Tau)
Description: Accumulation ratio of the analyte in plasma at steady state after multiple dose administration over a uniform dosing interval tau, expressed as ratio of AUC at steady state and after single dose
Time Frame: as for outcome 11
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 9
Ratio of AUC | 1.32 (23.4) | 1.11 (14.4) | 1.27 (18.1) | 1.49 (23.7) | 1.19 (18.6) | 1.42 (22.3) | 1.47 (32.8) | 1.21 (45.0)

ADVERSE EVENTS:
Time Frame: 4 days for SRD period + 17 days for MRD period
Groups:
- Placebo- Chinese: Matching placebo tablet: oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Chinese subjects
- Placebo- Japanese: Matching placebo tablet: oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Japanese subjects
- Placebo- Caucasian: Matching placebo tablet: oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Caucasian subjects
- BI 113608 - 10 mg - Chinese: 2 conventional tablets 5 mg BI 113608 oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 days (MRD period) in Chinese subjects
- BI 113608 - 10 mg - Japanese: 2 conventional tablets 5 mg BI 113608 oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Japanese subjects
- BI 113608 - 10 mg - Caucasian: 2 conventional tablets 5 mg BI 113608 oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Caucasian subjects
- BI 113608 - 25 mg - Chinese: 1 conventional tablet 25 mg BI 113608 oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Chinese subjects
- BI 113608 - 25 mg - Japanese: 1 conventional tablet 25 mg BI 113608 oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Japanese subjects
- BI 113608 - 50 mg - Chinese: 2 conventional tablets 25 mg BI 113608 oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Chinese subjects
- BI 113608 - 50 mg - Japanese: 2 conventional tablets 25 mg BI 113608 oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Japanese subjects
- BI 113608 - 50 mg - Caucasian: 2 conventional tablets 25 mg BI 113608 oral administration, single dose (SRD period) followed by twice a day for 13 days plus a single dose on day 14 (MRD period) in Caucasian subjects
Arm/Group | Placebo- Chinese | Placebo- Japanese | Placebo- Caucasian | BI 113608 - 10 mg - Chinese | BI 113608 - 10 mg - Japanese | BI 113608 - 10 mg - Caucasian | BI 113608 - 25 mg - Chinese | BI 113608 - 25 mg - Japanese | BI 113608 - 50 mg - Chinese | BI 113608 - 50 mg - Japanese | BI 113608 - 50 mg - Caucasian
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/7 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 3/9 | 5/7 | 5/9 | 2/9 | 9/9 | 7/9 | 4/9 | 9/9 | 7/9 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo- Chinese (N=9) | Placebo- Japanese (N=9) | Placebo- Caucasian (N=7) | BI 113608 - 10 mg - Chinese (N=9) | BI 113608 - 10 mg - Japanese (N=9) | BI 113608 - 10 mg - Caucasian (N=9) | BI 113608 - 25 mg - Chinese (N=9) | BI 113608 - 25 mg - Japanese (N=9) | BI 113608 - 50 mg - Chinese (N=9) | BI 113608 - 50 mg - Japanese (N=9) | BI 113608 - 50 mg - Caucasian (N=9)
Folliculitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 8 | 4 | 8
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Eyelid skin dryness (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 6
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal ulceration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.